CLINICAL TRIAL: NCT02224066
Title: Assessment of Platelet REACtivity After Transcatheter Aortic Valve Implantation
Brief Title: Platelet Reactivity After TAVI: A Multicenter Pilot Study
Acronym: REAC-TAVI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Meixoeiro (Other Government)
Responsible Party: Principal Investigator, Andres Iñiguez Romo, MD, PhD, Chief, Cardiology Department, Hospital Alvaro Cunqueiro, Hospital de Meixoeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEIX-VALV-002; REAC TAVI (Other: 201401)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Severe Aortic Valve Stenosis; Transcatheter Aortic Valve Implantation; Transcatheter Aortic Valve Replacement
Keywords: Aortic stenosis; TAVI; TAVR; Transcatheter aortic valve implantation; Ticagrelor; Antiplatelet reactivity
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Ticagrelor; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ticagrelor (Experimental): Patients with high-on-treatment platelet reactivity (PRU ≥ 208)
  Interventions: Drug: Ticagrelor 90 mg twice per day during three months following TAVI
- Aspirin/Clopidogrel (Active Comparator): Patients with high-on-treatment platelet reactivity (PRU ≥ 208)
  Interventions: Drug: Aspirin 100 mg plus Clopidogrel 75 mg daily during three months following TAVI
- Registry arm (No Intervention): Patients with normal-on-treatment platelet reactivity (PRU < 208) will continue with Aspirin 100 mg plus Clopidogrel 75 mg daily during three months following TAVI.

INTERVENTIONS:
Drug: Ticagrelor 90 mg twice per day during three months following TAVI
  Arms: Ticagrelor
Drug: Aspirin 100 mg plus Clopidogrel 75 mg daily during three months following TAVI
  Arms: Aspirin/Clopidogrel

SUMMARY:
A high platelet reactivity in patients with severe symptomatic Aortic Stenosis (AS) selected for TAVI (Transcatheter aortic valve implantation) procedure has been demonstrated previously, and the use of double antiaggregation therapy (DAPT) with Clopidogrel and Acetylsalicylic acid (ASA) do not achieve consistent and adequate suppression of platelet reactivity. The purpose of this study is evaluate the efficacy of ticagrelor alone versus DAPT with clopidogrel and aspirin for the suppression of high platelet reactivity following TAVI.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects should fulfill the following criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Adult patients (more than 18 years) with ability to understand and accept the participation in the clinical trial.
3. Patients with degenerative symptomatic severe AS accepted for TAVI after evaluation of the Heart Team of each center.
4. Patients who are not participating in any other clinical trial or research study (registries allowed).

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Recent stroke <14 days prior to TAVI, non-revascularized severe coronary or carotid artery disease (>70% stenosis) or life expectancy < 12 months
2. Patients under chronic oral anticoagulation
3. Patients with proven allergy to aspirin, clopidogrel or ticagrelor
4. Patients that after TAVI cannot undergo a regimen of single or dual antiplatelet therapy for 3 months due to a new post-TAVI medical indication
5. Known pregnancy or breast-feeding
6. Concomitant oral or intravenous therapy with potent inhibitors of cytochrome P450 3A (CYP3A) that cannot be suspended during the course of the study. Medications considered as potent inhibitors are: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin (or erythromycin but not astromicin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and more than a daily liter of grapefruit juice.
7. Thrombocytopenia (<50,000 platelets U/L) well documented and clinically relevant.
8. Patients with documented moderate or severe hepatic insufficiency
9. Any condition that may put the patient at risk or influence the outcome of the trial
10. Patients previously randomized in this trial or in another clinical trial with an investigational product or device over the past 30 days.
11. Patients who cannot attend follow up visits scheduled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of ticagrelor compared to clopidogrel and aspirin for the suppression of residual platelet reactivity by a system to verify the patient's platelet reactivity (VerifyNow P2Y12 assay). | Three months after antiplatelet treatment initiation following procedure.

SECONDARY OUTCOMES:
Evaluate the effectiveness of ticagrelor compared to clopidogrel and aspirin for the suppression of residual platelet reactivity by VerifyNow P2Y12 assay. | Six hours after antiplatelet treatment initiation following procedure.

OTHER OUTCOMES:
Assess the safety of antiplatelet monotherapy with ticagrelor compared to DAPT with aspirin and clopidogrel, with regard to the incidence of investigator-reported clinical events according to predefined criteria, including bleeding definitions. | Three months after antiplatelet treatment initiation following procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Iñiguez Romo, MD;Phd, Principal Investigator — Xerencia de Xestión Integrada de Vigo; Victor A Jimenez Diaz, MD; Msc, Principal Investigator — Xerencia de Xestión Integrada de Vigo; Pablo Juan Salvadores, Pharma; MPH, Study Director — Xerencia xestión integrada de Vigo
Locations (7):
- Spain (7):
  - Hospital Clinic Universitari Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Santa Creu i Sant Creu, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Ussia GP, Scarabelli M, Mule M, Barbanti M, Sarkar K, Cammalleri V, Imme S, Aruta P, Pistritto AM, Gulino S, Deste W, Capodanno D, Tamburino C. Dual antiplatelet therapy versus aspirin alone in patients undergoing transcatheter aortic valve implantation. Am J Cardiol. 2011 Dec 15;108(12):1772-6. doi: 10.1016/j.amjcard.2011.07.049. Epub 2011 Sep 10. PMID 21907949
- [Background] Makkar RR, Fontana GP, Jilaihawi H, Kapadia S, Pichard AD, Douglas PS, Thourani VH, Babaliaros VC, Webb JG, Herrmann HC, Bavaria JE, Kodali S, Brown DL, Bowers B, Dewey TM, Svensson LG, Tuzcu M, Moses JW, Williams MR, Siegel RJ, Akin JJ, Anderson WN, Pocock S, Smith CR, Leon MB; PARTNER Trial Investigators. Transcatheter aortic-valve replacement for inoperable severe aortic stenosis. N Engl J Med. 2012 May 3;366(18):1696-704. doi: 10.1056/NEJMoa1202277. Epub 2012 Mar 26. PMID 22443478
- [Background] Tousek P, Kocka V, Sulzenko J, Bednar F, Linkova H, Widimsky P. Pharmacodynamic effect of clopidogrel in patients undergoing transcatheter aortic valve implantation. Biomed Res Int. 2013;2013:386074. doi: 10.1155/2013/386074. Epub 2013 Jul 15. PMID 23956980
- [Background] Price MJ, Angiolillo DJ, Teirstein PS, Lillie E, Manoukian SV, Berger PB, Tanguay JF, Cannon CP, Topol EJ. Platelet reactivity and cardiovascular outcomes after percutaneous coronary intervention: a time-dependent analysis of the Gauging Responsiveness with a VerifyNow P2Y12 assay: Impact on Thrombosis and Safety (GRAVITAS) trial. Circulation. 2011 Sep 6;124(10):1132-7. doi: 10.1161/CIRCULATIONAHA.111.029165. Epub 2011 Aug 29. PMID 21875913
- [Background] Husted S, James S, Becker RC, Horrow J, Katus H, Storey RF, Cannon CP, Heras M, Lopes RD, Morais J, Mahaffey KW, Bach RG, Wojdyla D, Wallentin L; PLATO study group. Ticagrelor versus clopidogrel in elderly patients with acute coronary syndromes: a substudy from the prospective randomized PLATelet inhibition and patient Outcomes (PLATO) trial. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):680-8. doi: 10.1161/CIRCOUTCOMES.111.964395. PMID 22991347
- [Derived] Jimenez Diaz VA, Tello-Montoliu A, Moreno R, Cruz Gonzalez I, Baz Alonso JA, Romaguera R, Molina Navarro E, Juan Salvadores P, Paredes Galan E, De Miguel Castro A, Bastos Fernandez G, Ortiz Saez A, Fernandez Barbeira S, Raposeiras Roubin S, Ocampo Miguez J, Serra Penaranda A, Valdes Chavarri M, Cequier Fillat A, Calvo Iglesias F, Iniguez Romo A. Assessment of Platelet REACtivity After Transcatheter Aortic Valve Replacement: The REAC-TAVI Trial. JACC Cardiovasc Interv. 2019 Jan 14;12(1):22-32. doi: 10.1016/j.jcin.2018.10.005. PMID 30621974